CLINICAL TRIAL: NCT00415974
Title: PACE-PC: Primary Care Management of Adolescent Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Kevin Patrick, MD, MS, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01CA121300-01 (NIH)
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: Obesity; Overweight; Weight Loss
Keywords: Weight Loss; Obesity; Overweight; Physical Activity; Nutrition; Primary Care Physicians; Primary Care; Counseling; Adolescent
MeSH Terms: conditions — Obesity; Overweight; Weight Loss; Motor Activity | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Usual Care (Other): Enhanced Usual Care Arm: This group will receive 2 face-to-face sessions with a health educator for dietary and health counseling in addition to an initial physician-patient visit. Educational materials that a patient might receive at his/her physician's office will also be provided at the initial health educator visit and monthly thereafter. This condition is called "Enhanced Standard Care" because it is, in fact, more than most obese adolescents currently receive in primary care offices in San Diego.
  Interventions: Behavioral: Physician Counseling; Behavioral: Health Educator; Behavioral: Health promotion materials on physical activity and nutrition
- Stepped Care (Experimental): PACE-PC is a 1-year stepped-care intervention (subdivided into three 4-month blocks) utilizing multiple modalities including clinician and tailored health educator counseling, phone counseling, mailed content for overweight adolescents and their family to promote improved diet and physical activity behaviors aimed at weight loss and weight loss maintenance.
  PACE-PC is designed to be based in the primary care setting and promotes involvement, management, and decision-making by the primary care provider about the level of PACE-PC step for each enrolled patient
  Participants randomized to the PACE-PC condition will be enrolled in Step 1 (the most intensive) for the first 4 months. Depending upon response at the end of Step 1, for the next 4 months adolescents will be triaged to Step 2 (less intensive) or will repeat Step 1. At 8 months, again based upon treatment response, triage will occur to either Step 3 (least intensive) or repetition of the previous step.
  Interventions: Behavioral: Physician Counseling; Behavioral: Health Educator; Behavioral: Phone Counseling; Behavioral: Health promotion materials on physical activity and nutrition

INTERVENTIONS:
Behavioral: Physician Counseling — Physician-patient visits will occur in the primary care setting and are scheduled at study onset (beginning of step 1) and at the end of the first year. An extra physician visit will occur for patients who do not progress from step 1 after two attempts. At study entry, physicians will discuss the purpose and importance of the intervention and encourage participation. Physicians will underline the value of attending all study visits and complying with study protocol and instructions. Subsequent physician visits will focus on weight loss progress and overcoming barriers.
Behavioral: Health Educator — Health education sessions are held with teens and parents at the primary care setting. These include information on nutrition, physical activity, and weight loss. Behavioral approaches are used to enhance the home environment, food preparation, and planned physical activity to elicit weight loss, including discovery of perceived and actual barriers to modification of eating and physical activity behaviors. The Health Educator focuses on problem-solving and tailored selection of behavior change skills to help participants overcome difficulties. In addition to reviewing the assessment and generating solutions to barriers, sample meal plans (including strategies for restricting calories) and pedometers will be distributed at the initial health educator visit. Pedometers are encouraged to monitor progress with physical activity goals. An initial binder is distributed to teen and parent participants at the initial session and subsequent materials are added with each visit.
Behavioral: Phone Counseling — Brief counseling calls will occur between PACE-PC participants and assigned counselors during all steps. In general, these calls occur on a bi-weekly to monthly basis in steps 1 and 2, and monthly in step 3. Such calls are intended to encourage continued goal attainment and progression and to promote healthy eating and physical activity behaviors. Counselors will review progress since the last clinical interaction (e.g., health educator visit, phone call, or physician visit) and help adolescents set new goals that are appropriate and attainable. Data from pedometers may be discussed during these sessions as an interim assessment of progress on physical activity behaviors between formal study measurement visits. After speaking with the adolescent, the counselor will talk with the parent (when feasible) to reinforce parental involvement and emphasize the importance of the healthy changes in the home environment to encourage goal attainment.
  Arms: Stepped Care
Behavioral: Health promotion materials on physical activity and nutrition — PACE-PC adolescents and their families will receive information regarding healthy eating and physical activity behaviors on a weekly basis via mail. These behavioral-based materials will educate participants and their families on healthy behaviors that are necessary for successful weight management. Topics will coincide with the intervention goals and include supplemental information to enhance quality of life and improve body image. Topics will include realistic goal-setting and attainment, how to handle holidays and celebrations, eating fast food, grocery shopping and food preparation, and relapse prevention, etc.. Topics will include specific strategies related to the adolescent's readiness to change to reflect processes that are most appropriate. Content from these materials will be addressed by the phone counselors to ensure that participants received and understood intervention messages.

SUMMARY:
This 12-month randomized controlled trial, sponsored by NIH/NCI, aims to reduce BMI in obese adolescents (ages 11 -13) by intervening on physical activity and nutrition behaviors within primary care settings.

PACE-PC is a theory-based stepped care program that enables pediatricians and primary care providers to intervene with obese adolescents to improve their anthropometric, metabolic, physiological, behavioral, and quality of life outcomes over a one-year period. The program integrates clinician counseling, health educator counseling, and phone and mail contact. It supports tailoring to the needs of obese adolescents and family members and promotes improved diet and physical activity behaviors, weight loss, and ultimately weight loss maintenance.

Participants will be randomly assigned to the Enhanced Usual Care or the PACE-PC stepped care condition. The Enhanced Standard Care condition includes an initial visit and counseling by a physician, 3 visits with a health educator, and materials on how to improve weight related behaviors.

The PACE-PC Stepped Care condition includes 3 steps (each lasting 4 months), with the first step being the most intensive:

Step 1 includes: a physician visit, monthly health educator visits, biweekly phone counseling, and weekly dissemination of nutrition and physical activity information

Step 2 includes: a health educator visits every other month, biweekly phone counseling, and weekly dissemination of nutrition and physical activity information

Step 3 includes: monthly phone counseling and weekly dissemination of nutrition and physical activity information

Participants randomized to the PACE-PC condition will be enrolled in Step 1 (the most intensive) for the first 4 months. Depending upon response at the end of Step 1, for the next 4 months adolescents will be triaged to Step 2 (less intensive) or will repeat Step 1. At 8 months, again based upon treatment response, triage will occur to either Step 3 (least intensive) or repetition of the previous step.

DETAILED DESCRIPTION:
Obesity in adolescence is becoming increasingly prevalent. Thirty years ago the prevalence of obesity among adolescents aged 12-19 years was approximately 6%. Between 1980 and 1994, the number of children and adolescents meeting criteria for overweight/obese, as defined by a body mass index (BMI) > 95% for children of the same age and gender, increased by 100% in the United States (Ogden, Flegal, Carroll et al., 2002). The increased prevalence of childhood obesity has been universal in all age, gender, and ethnicity classification. As of the year 2002, over 16% of adolescents are obese in the United States (Ogden et al., 2002) and this problem is even more important in selected regions of the country. For example, the California Center for Public Health Advocacy, (2002), reported that the percentage of 5th, 7th, and 9th graders (ages 10 and 15 years) who had a body mass index (BMI) greater than the 95th percentile ranged from 17.3% - 36% depending upon school attended. Overall childhood obesity is increasingly recognized as one of the nation's most important health issues (IOM, 2004).

Obesity affects all parts of the body including the brain, lungs, heart, liver, pancreas, intestines, kidneys, and skeleton. Consequently, children who meet the criteria for obesity are at risk for serious health problems. A lower quality of life has also been shown among children who are overweight (Schwimmer et al., 2003). Adolescent obesity is also a significant predictor of adult obesity (Clark & Lauer, 1993; Mossberg, 1989). Approximately 1/3 of overweight adults are overweight before 20 years of age. An even larger percentage of morbidly obese adults became obese as children (Rimm & Rimm, 1976). Overweight adolescents are the pediatric group carrying the highest risk for childhood obesity persistence into adulthood (Whitaker et al., 1997).

There is strong evidence of the health benefits of physical activity (USDHHS, 1996; Biddle et al., 2004) including improvements in risk of cancer, longevity, cardiovascular diseases, (CVD), CVD risk factors, diabetes, obesity, osteoporosis, immune functioning, and mental health. More recent guidelines from the Dietary Guidelines for Americans (USDHHS, 2005) and the United Kingdom Health Education Authority recommend 60 minutes of daily PA for youth (Biddle et al., 1998; Cavill et al., 2001). Although national survey data in the U.S. indicate that about two-thirds of adolescent boys and about one-half of adolescent girls are meeting an adult-oriented recommendation for vigorous activity (Pate et al., 1994), objective measures suggest less than 40% of teens are meeting the 60 minute guideline (Pate et al., 2002). Females, older adolescents, minorities and disadvantaged youth are even less likely to be meeting this recommendation (USDHHS, 1998).

Poor dietary behaviors are a known risk factor for the development of obesity, as well as for the nation's three leading causes of death: CHD, cancer and stroke. Research supports that a diet rich in fruits and vegetables and low in fat is important in preventing these chronic diseases, and is recommended by the USDA, USDHHS, Surgeon General, NRC, NHLBI, NCI, ACS, and AHA (USDA, 1991; USDA, 1992; National Research Council, 1989; NHLBI, 1990; NHLBI, 1991; NCI, 1991; Weinhouse et al., 1991; AHA, 1988). Although national surveys indicate a decline in the average proportion of calories from total and saturated fat over the past several decades, the CDC estimated in 2000 that only 38% of individuals 2 years and older met the recommendation for total fat intake and 41% of these individuals met the recommendation for saturated fat intake. Simple dietary restriction has not been associated with successful weight control (NAS, 1991) and may even result in a nutritionally inadequate diet. Thus, rather than focusing only on limiting total energy intake, it is important to promote a diet that is nutrient dense: high in vegetables, fruits, grains, and other fiber-rich plant foods, yet low in fat, at a given level of energy intake.

Obesity is a chronic health condition (WHO, 1998). As such, long-term medical management is appropriate, with particular attention to comorbidity development and identification. According to the Institute of Medicine (IOM), primary care is "the provision of integrated, accessible healthcare services by clinicians who are accountable for addressing a large majority of personal healthcare needs, developing a sustained partnership with patients and practicing within the context of family and community" (IOM, 1996)." Various studies have evaluated primary healthcare and found that primary care provides accessible, comprehensive, coordinated, adequately communicated, longitudinal healthcare (Flocke, 1997; Safran et al., 1998; Starfield, 1998). Primary healthcare has been called the "medical home;" and the American Academy of Pediatrics (AAP) (1992, p. 251) describes the "medical home" (with respect to care for infants, children, and adolescents) as: "accessible, continuous, comprehensive, family centered, coordinated, and compassionate"; "delivered or directed by physicians who are able to manage or facilitate essentially all aspects of pediatric care"; and involving physicians who "should be known to the child and family and able to develop a relationship of mutual responsibility and trust." Thus, pediatricians, family physicians and others in primary care have many opportunities to assist with obesity treatment in children.

Although children and adolescents visit physicians less often than other age groups, the amount of contact is extensive. Overweight youth may be even more likely to visit their primary care physician as compared to non-overweight children (Gauthier et al., 2000). In addition, adolescents have indicated a willingness and desire to discuss weight issues with their healthcare provider (Hodgson et al., 1986; Marks et al., 1983).

The American Heart Association and the American Diabetes Association advocate primary care counseling for modifiable coronary artery disease risk factors, including obesity, during preventive health examinations (ADA, 2001; Grundy et al., 1997). In a recent study conducted in two primary care practices in Louisiana (Huang et al., 2004), primary care practitioner counseling on weight loss was well-received by patients and effective in increasing patients' understanding of the negative health impact of obesity. However, also identified in this study was the lack of sufficient guidance on weight management strategies for primary care practitioners. Potential reasons for this deficiency include: insufficient physician confidence, knowledge and counseling skills, as well as lack of time, resources and under use of dietitians contribute to inadequate counseling on diet, physical activity, and weight loss (Yeager et al., 1996) The extent and content of physician counseling about diet, exercise, and weight loss are inadequate (Galuska et al., 1999; Nawaz et al., 2000). This is discouraging given the fact that physician-patient interactions regarding healthy diet habits have been shown to effect change resulting in improved eating habits (USPSTF, 2002) and weight loss (Nawaz, 2000).

Given its potential, it is surprising how little research has been conducted on primary care interventions for obesity in childhood. To our knowledge, a study by Saelens et al., 200 is the only study to date evaluating a primary care-based behavioral therapy program for weight control management in adolescents. One pilot study evaluates the feasibility of introducing a low glycemic index diet at the primary care setting as a primary-care-based therapy (Young et al., 2004). While preliminary data are promising, this treatment only addresses nutritional issues associated with obesity.

The stepped care treatment scheme for chronic disease has been advocated for some time (Black et al., 1984; Brownell, 1992). Usually this strategy is a step-up one with the least intensive, least expensive, and least dangerous approach used first with all individuals. Only non-responders progress to the next most intensive step, followed by additional increases in intervention intensity if subjects fail to respond.

While most stepped care approaches are modeled after the above-described step-up method, the current model advocated by the United States Preventive Services Task Force (USPSTF) and the NHLBI adheres to a step-down approach where all patients begin with the most intensive step followed by less intensive interactions as patients gain self-efficacy and self-management skills. In the USPSTF review of 17 randomized controlled trials of high-intensity (more than monthly face-to-face contact), medium-intensity (monthly face-to-face contact), and low-intensity (less than monthly interpersonal contact) interventions for obesity (McTigue et al., 2003), the most effective treatment methods were of high intensity which combined two to three components (nutrition education, diet and exercise counseling, and behavioral strategies) within the first 3 months of therapy. These methods were able to achieve weight loss ranges from 3 to 5 kilograms at the one year follow-up visit. In addition, the NHLBI obesity management recommendations (NHLBI, 2000) encourage regular and frequent medical follow-up in the first 6 months of therapy followed by a tapered visit frequency schedule. Weight management is an important principle emphasized by the NHLBI, which encourages continued therapeutic modalities during this "maintenance period" (which may continue indefinitely) to prevent regain of weight lost. Structured treatment programs with regular follow-up improve long-term weight loss and maintenance (Perri et al., 1993; Lantz et al., 2003).

Research to date suggests that a primary care-based "stepped-down" care model is palatable and may be efficacious in promoting weight loss on a population scale.

In sum, the proposed study will help fill several gaps in the literature: There is very little known about:

* How to enable primary care pediatricians, family physicians and others in "front line" clinical settings to successfully intervene with their obese adolescent patients. In many geographical areas alternative interventions for adolescent obesity (e.g., specialist care or community-based programs) might either be non-existent or difficult to access. Thus the role of primary care clinicians may be even more important.
* Obesity interventions of any type for individuals under the age of 18 years. The increase in the prevalence of this health problem is far outstripping medical knowledge regarding treatment in this population.
* The impact of an intervention like PACE-PC on anthropometric, metabolic, physiological and behavioral measures and outcomes in obese adolescents. Understanding how interventions do-and do not-alter key health related factors associated with obesity is critical to the overall field of pediatric obesity.
* Whether adherence to, and outcomes associated with, obesity treatment can be improved through a multi-channel, stepped care program like PACE-PC. There are no reports in the literature of stepped care approaches to pediatric obesity, especially those that incorporate elements of the chronic care model.
* Whether weight change brought about by one year of a multimodal intervention can be sustained for an additional year through a less intensive maintenance intervention. Maintenance of weight status following weight loss is very difficult. Exploring methods to accomplish this is important.
* The cost-effectiveness of interventions such as PACE-PC for obese adolescents. If this intervention is to become generalized, someone must be willing to pay for it, either employers or other entities at risk for healthcare expenses, or consumers themselves. Increased knowledge about the cost effectiveness of PACE-PC will inform decisions made by these parties.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females, ages 11-13 who are obese (> 95% Body Mass Index for age and gender). Participants must have:

  * a home telephone and permanent residence with the intent to stay in the San Diego area over the entire study period;
  * willingness to return to the pediatrician for counseling sessions;
  * ability to attend measurement visits at the PACE research office.

Exclusion Criteria:

* Any prospective participant with any comorbidities of obesity that require immediate sub-specialist referral including pseudotumor cerebri, sleep apnea, obesity hypoventilation syndrome, and orthopedic problems will be excluded from the study.
* Additionally, participants will also be excluded if they are over 285 pounds (limits of DXA machine), have any pulmonary, cardiovascular or musculoskeletal problem that would limit ability to comply with moderate-level physical activity (e.g. walking), have a history of substance abuse, or other psychiatric disorder that would impair compliance with the study protocol, or are using any medications which alter body weight.
* Patients in foster care will be ineligible due to difficulty in obtaining follow-up measures should they move from home to home.

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Primary: The primary outcome of this study is to compare at 12 months, the effects of the PACE-PC intervention and enhanced standard care on BMI z-score among obese (> 95 percentile for age) male and female adolescents aged 11 -13. | baseline, 4 months, 8 months, 12 months

SECONDARY OUTCOMES:
Secondary: Secondary outcomes will be: 1) anthropometric measures (BMI, waist circumference, body fat); 2) metabolic and physiological manifestations of obesity (fasting insulin, fasting blood glucose and blood lipid levels); 3) behavioral measurement | baseline, 4 mos, 8 mos, 12 mos

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Patrick, MD, MS, Principal Investigator — UCSD
Locations (1):
- UCSD - CALIT2- Atkinson Hall, La Jolla, California, United States

REFERENCES:
- [Derived] Kolodziejczyk JK, Gutzmer K, Wright SM, Arredondo EM, Hill L, Patrick K, Huang JS, Gottschalk M, Norman GJ. Influence of specific individual and environmental variables on the relationship between body mass index and health-related quality of life in overweight and obese adolescents. Qual Life Res. 2015 Jan;24(1):251-61. doi: 10.1007/s11136-014-0745-1. Epub 2014 Jul 1. PMID 24980678